CLINICAL TRIAL: NCT06663696
Title: Evaluation of the Safety and Clinical Performance of the Biodegradable Polymer-Coated Sirolimus-Eluting Stent in All-Comer Patients With Multivessel Coronary Artery Disease
Brief Title: CRUZ Tunisia-Multivessel Registry
Status: Recruiting | Type: Observational
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CRUZ/TUNISIA-MV/01-2023
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Patient Population With Multivessel Disease
Keywords: Multivessel disease, Supraflex Cruz, SES

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population with multivessel disease: Supraflex Cruz Sirolimus-eluting Coronary Stent System
  Interventions: Device: Supraflex Cruz Sirolimus-eluting Coronary Stent System

INTERVENTIONS:
Device: Supraflex Cruz Sirolimus-eluting Coronary Stent System — Biodegradable polymer-coated, cobalt-chromium sirolimus-eluting coronary stent

SUMMARY:
The primary objective of this registry is to evaluate the safety and clinical performance of the biodegradable polymer-coated Supraflex Cruz Sirolimus-eluting Stent (SES) in an unselected, all-comer patient population with multivessel disease. This population represents daily clinical practice and includes patients requiring coronary revascularization with drug-eluting stents (DES).

DETAILED DESCRIPTION:
This is a prospective, observational, single-arm, multi-center, registry designed to evaluate the safety and clinical performance of the Supraflex Cruz SES in an unselected, all-comer patient population with multivessel disease. The multivessel disease, defined as the presence of two or more vessels that will be exclusively treated with the Supraflex Cruz SES. The registry aims to reflect daily clinical practice including, but not limited to patients with chronic coronary artery disease (CAD) as well as acute coronary syndrome (STEMI and NSTEMI).

All patients will be followed as per routine clinical practice together with either telephonic or clinical follow-up at 30 days, 6 months, and 12 months after the index procedure.

Subgroups are pre-specified for post-hoc exploratory analyses with respect to the primary endpoint of Target Lesion Failure (TLF) at 12 months. The following subgroups are pre-defined according to their presentation at enrolment:

1. Treatment in relation to clinical presentation [Acute Coronary Syndrome (ACS)]
2. Treatment in relation to specific lesion subsets [Left Main, Chronic Total Occlusion]
3. Patients undergoing atherectomy

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age
2. Patients with symptomatic coronary artery multivessel disease requiring the implantation of at least two Supraflex Cruz stents into the coronary vasculature during the index procedure
3. The patient, or legal representative, has been informed of the nature of the registry and has consented to participate and authorised the collection and release of his/her medical information by signing a Patient Informed Consent Form
4. The patient is willing and able to co-operate with study procedures and required follow up visits

Exclusion Criteria:

1. Women with known pregnancy or who are lactating
2. High probability of non-adherence to the follow-up requirements (due to social, psychological, or medical reasons)
3. Currently participating in another study that has not completed the primary endpoint or that clinically interferes with the current registry requirements
4. Patients has a known hypersensitivity or contraindication to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI, cobalt chromium, sirolimus or contrast media

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population with multivessel disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  TLF is defined as: "a composite endpoint of cardiovascular death, target vessel myocardial infarction (TV-MI), or clinically driven target lesion revascularization (CD-TLR)".

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | 30 days, 6 months
All-cause mortality | 30 days, 6 months, and 12 months
Any myocardial infarction (MI), includes non-target vessel territory | 30 days, 6 months, and 12 months
Any revascularization | 30 days, 6 months, and 12 months
Definite/probable stent thrombosis | 30 days, 6 months, and 12 months
Target Vessel Failure (TVF) | 30 days, 6 months, and 12 months
  TVF is defined as: "a composite endpoint of cardiovascular death, target vessel myocardial infarction, or clinically driven target vessel revascularization"

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Nadhem HAJLAOUI, Principal Investigator — University of Tunis El Manar, Tunisia
Locations (2):
- Tunisia (2):
  - Sahloul Hospital, Sousse
  - Habib Thameur Hospital, Tunis

IPD SHARING:
Plan to Share IPD: No